CLINICAL TRIAL: NCT04128800
Title: A Single-center, Single-arm Exploratory Clinical Study of Apatinib Mesylate Tablets Combined With S-1 in the Treatment of Second-line or More Advanced Small Cell Lung Cancer
Brief Title: Appatinib Combined With S-1 in the Treatment of Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AHEAD-HBH
Record Dates: First submitted 2019-10-15; First posted 2019-10-16 (Actual); Last update posted 2019-10-16 (Actual); Status verified 2019-10

CONDITIONS: Small Cell Lung Cancer
Keywords: apatinib S-1; Advanced lung cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Apatinib and S-1 group (Experimental)
  Interventions: Drug: Apatinib S-1

INTERVENTIONS:
Drug: Apatinib S-1 — apatinib 250 mg PO qd; S-1 40 mg PO in the morning and 60 mg PO in the evening; 14 days in combination, 21 days in a cycle.
  Other Names: apatinib mesylate tablets

SUMMARY:
To evaluate the objective remission rate and disease control rate of apatinib mesylate tablets combined with S-1 in the treatment of advanced small cell lung cancer patients with failed or dangerous radiotherapy or chemotherapy

DETAILED DESCRIPTION:
Lung cancer is one of the malignant tumors with the highest morbidity and mortality in the world. Small cell lung cancer accounts for about 15-20% of all lung cancer. Although the initial treatment is sensitive to radiotherapy and chemotherapy, patients with small cell lung cancer are prone to recurrence and metastasis in the early stage, and ultimately lead to death due to the lack of effective treatment after the disease progresses. Patients with relapsed small cell lung cancer had a poor prognosis; untreated patients had only two to three months of expected survival.Therefore, it is urgent to find a method to treat SCLC.

Two single-arm phase II clinical studies on small cell lung cancer have evaluated the efficacy and safety of bevacizumab combined with first-line chemotherapy for extensive SCLC. Two phase II single arm studies showed good efficacy and safety. Apatinib and bevacizumab are both antiangiogenic agents. S-1 is a new oral fluoropyrimidine anticancer agent, but S-1 has shown a high remission rate for metastatic NSCLC and relapsed NSCLC.

In view of the good efficacy and tolerability of oral chemotherapeutic agent S-1, and the lack of suitable targeted drugs after NGS treatment in relapsed S LCL patients after previous multithreaded treatment, this clinical trial is to study the efficacy and safety of combination of anti-angiogenesis drugs and S-1 in patients with failed or dangerous SCLC after second-line or more radiotherapy and chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. The informed consent of the patient must be obtained before any research steps are carried out.
2. Confirmation of SCLC: Histological diagnosis or two imaging diagnoses must be made.
3. Late stage of SCLC, failure of second-line radiotherapy and chemotherapy or dangerous type of patients
4. Male or female subjects > 18 years old, < 75 years old
5. There are objective lesions that can be measured by CT.
6. The activity status of KPS was above 80 points.
7. Within 14 days before admission, the bone marrow, liver and kidney functions detected by the central laboratory should meet the following laboratory data requirements:

   Hemoglobin ≥ 9.0 g/dl; absolute neutrophil count (ANC)1,500 /mm3 ; platelet count ≥ 50,000 /ul; total bilirubin < 2 mg/dL (3 mg/dL, Child B); ALT and AST < 5-fold normal value upper limit; alkaline phosphatase < 4-fold normal value upper limit; PT > 50% or PT-INR < 2.3, or greater than the control value < 6 seconds.
8. For subjects taking warfarin, the subjects were closely monitored at least once a week until the INR measurement of the subjects was stable at the time of each administration according to the local treatment standards.
9. The upper limit of normal serum creatinine < 1.5 times is
10. For pregnant women, the results of serum pregnancy test must be negative within 14 days before the start of treatment.
11. All male and female patients participating in this study must adopt reliable contraceptive measures during the trial and within two week.

Exclusion Criteria:

1. KPS < 60 points, or expected survival < 3 months.
2. Severe cardiovascular diseases .
3. Uncontrollable hypertension .
4. History of human immunodeficiency virus (HIV) infection .
5. Active clinical severe infections (Grade 2, NCI-CTCAE Version 3.0) .
6. Epilepsy patients requiring medication (e.g. steroids or antiepileptic drugs) .
7. History of allogeneic organ transplantation .
8. Patients with signs of hemorrhage or history of disease.
9. Patients undergoing renal dialysis.
10. Chronic obstructive pulmonary emphysema .
11. Gastrointestinal bleeding within 30 days before admission .
12. Patients have a history of esophageal varices bleeding, and subsequently did not receive effective treatment or treatment to prevent recurrence of bleeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-10 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate(ORR) | one year

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | one year

OTHER OUTCOMES:
Progression free survival (PFS) | one year
Overall survival (OS) | one year
Quality of life (QoL) | one year

CONTACTS AND LOCATIONS:
Overall Officials: Ning bo Liu, MD, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code